CLINICAL TRIAL: NCT06268678
Title: The Effect of Menstrual Cycle Phase on Muscle Protein Synthesis Following Protein Ingestion and Resistance Exercise in Young Women
Brief Title: The Effect of Menstrual Cycle Phase on Muscle Protein Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Pvolve (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 4539513
Record Dates: First submitted 2024-01-10; First posted 2024-02-20 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Menstrual Cycle Phase; Muscle Protein Synthesis

STUDY DESIGN:
Intervention Model Description: Randomised cross-over design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follicular (Experimental): Follicular phase assessment of muscle protein synthesis.
  Interventions: Other: Phase of the menstrual cycle
- Luteal (Experimental): Luteal phase assessment of muscle protein synthesis
  Interventions: Other: Phase of the menstrual cycle

INTERVENTIONS:
Other: Phase of the menstrual cycle — Follicular or luteal phase

SUMMARY:
The combination of dietary protein ingestion and resistance exercise are essential to increase muscle protein synthesis. The vast majority of studies assessing protein intake following resistance exercise in young adults has been conducted exclusively in men or in studies where both men and women are assessed. The increase in muscle mass is thought to be impacted by sex hormones that fluctuate across different phases of the menstrual cycle. However, the effect of menstrual cycle phase on muscle protein synthesis following exercise is not known.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-40 years
* BMI between 18 and 30 kg/m2
* Recreationally active
* Regular menstrual cycle

Exclusion Criteria:

* Smoking or use of tobacco containing products
* Irregular menstrual cycle
* Currently on any form of hormonal contraception
* Post-menopausal
* Pregnant or breastfeeding
* Diagnosed metabolic/pulmonary/musculoskeletal illness
* Diagnosed cardiovascular disease or hypertension
* Use of medications that may impact protein metabolism or are anti-inflammatory
* Gastrointestinal disorders
* Allergy to pomegranate or amino acids
* Injuries that would impact ability to complete study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-09-28 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | 7 hours
  The rate of synthesis of new muscle protein

SECONDARY OUTCOMES:
Plasma amino acid kinetics | 7 hours
  The appearance of amino acids in the circulation.
Serum insulin concentrations | 7 hours
  Basal and postprandial concentrations of serum insulin
Sex hormone concentrations | 5 minutes
  Serum oestrogen and progesterone
Energy expenditure | 20 minutes
  Basal metabolic rate

CONTACTS AND LOCATIONS:
Overall Officials: Francis Stephens, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No